CLINICAL TRIAL: NCT01099956
Title: Low Grade Inflammation in Type 1 Diabetes Children
Acronym: Coccinelle
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2009/28
Record Dates: First submitted 2010-03-22; First posted 2010-04-08 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Type 1 Diabetes; Inflammation
Keywords: type 1 diabetes; children; low grade inflammation; cytokine; CRP
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- diabetes group
- control group

SUMMARY:
The study propose to measure the inflammation level in type 1 diabetes children with the cytokine analysis compared to non diabetic children of the same sibling and to healthy children.

DETAILED DESCRIPTION:
The increase of type 1 diabetes incidence, particularly in young children leads to conduce new diagnostic and therapeutic strategies, notably for associated chronic morbidity.Measurement of chronic inflammation, with modification of the balance between pro-inflammatory cytokines and anti-inflammatory cytokines, could lead to detect patients with high risk to diabetes chronic morbidity.

After parental consent, blood sampling will be carried out by micromethod for cytokine (500 µl) and CRPhs dosages and glycemia (100 µl) and glycated hemoglobin (1 µl). Urine will be collected (50 ml) in the morning for further researches.

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetes children group :

* Children aged 2 to 17 years
* Type 1 diabetes children

Controlled group :

* Children aged 2 to 17 years
* Brother or sister of type 1 diabetes children

Exclusion Criteria:

* Per os or inhaled corticoid in the previous month of inclusion
* Acute infectious disease in the previous week of inclusion
* Other chronic disease than diabetes type1

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 60 children in type 1 diabetes group and 30 children in control group
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Increase of Interleukine 6 in group DTI versus control group | Once at inclusion

SECONDARY OUTCOMES:
Increase of others cytokines (IL1-beta, l'IL-4, l'IL-10 and TNF alpha) and increase of High sensitivity CRP in group DTI versus control group | Once at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pascal BARAT, MD, Principal Investigator — University Hospital, Bordeaux, France
Locations (1):
- Children Hospital, Endocrinology Unit, Bordeaux, France